CLINICAL TRIAL: NCT04675762
Title: A Randomised Controlled Trial of Combinating an Immune Modulator Fingolimod With Alteplase Bridging With Mechanical Thrombectomy in Acute Ischemic Stroke
Brief Title: Combinating Fingolimod With Alteplase Bridging With Thrombectomy in Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huizhou Municipal Central Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jinhua Center Hospital (Unknown); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMMUTAS
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Inflammation
Keywords: Fingolimod Hydrochloride; Intravenous thrombolysis; Mechanical thrombectomy; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Inflammation; Ischemic Stroke | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fingolimod with standard therapy (Experimental): Patients will be treated with standard alteplase bridging and mechanical thrombectomy with fingolimod.
  Interventions: Drug: Fingolimod
- Placebo with standard therapy (Placebo Comparator): Patients will be treated with standard alteplase bridging and mechanical thrombectomy with placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fingolimod — Patients randomized to fingolimod will also receive fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is about one hour prior to mechanical thrombectomy.
  Arms: fingolimod with standard therapy
Other: Placebo — Patients randomized to fingolimod will also receive placebo once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is about one hour prior to mechanical thrombectomy.
  Arms: Placebo with standard therapy

SUMMARY:
Proof-of concept clinical trials have indicated that the sphingosine-1-phosphate receptor modulator fingolimod may be efficacious in attenuating brain inflammation and improving clinical outcomes in patients with AIS as a single therapy beyond 4.5 hours of disease onset, or in combination with alteplase within 4.5 hours of disease onset. So in this study the investigators try to determine whether the addition of fingolimod, administered within 24 hours after the onset of symptoms in patients receiving alteplase bridging with mechanical thrombectomy, improves radiologic and clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled design clinical trial, in multiple stroke centers of China. The total sample size will be 118. Patients being treated with standard alteplase bridging and mechanical thrombectomy will be randomly assigned in a 1:1 ratio to receive fingolimod or placebo.

Patients aged between 18 and 85 with anterior circulation AIS who are eligible for alteplase and mechanical thrombectomy commenced within 24 hours of stroke onset or awakening with stroke (if within 24 hours from the midpoint of sleep) will be enrolled if they present with an infarct core volume ≤ 100 mL and penumbra ≥ 15 mL with at least 20% mismatch (as evaluated by CTP) and intracranial occlusion in proximal cerebral arteries. Exclusion criteria are (1) pre-existing neurologic disability (a score greater than 2 on the mRS); (2) contraindication of fingolimod.

As standard care, all patients will receive standard dose intravenous alteplase (0.9 mg per kilogram, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg) and mechanical thrombectomy delivered at the site of intracranial vessel occlusion. Patients randomized to fingolimod group or placebo group will receive fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg or placebo once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is about one hour prior to mechanical thrombectomy.

The kinetics of lymphocyte subset alteration will be monitored in whole-blood samples from all fingolimod- treated patients at the baseline, which will precede the first dose, day 1 and day 7. Mononuclear cells will be isolated from the whole-blood specimens and stained with antibodies to CD4-FITC, CD8-PE, CD19-PerCP, CD56-PE (BD Biosciences, Franklin Lakes, NJ, USA). Data will be acquired using a FACS Caliber (Becton Dickinson Immunocytometry Systems, San Jose, CA, USA) and analyzed with Flow Jo software (Tree Star, Ashland, OR, USA).

The primary outcome is the ratio of mRS 0-2 (%) at 90 day. Secondary outcomes are the salvaged ischemic tissue index (%) from baseline to 7 day, the growth in infarct volume (mL) from 24 hour to 7 day, the penumbral salvage volume (mL) from baseline to 1 day, the frequency of parenchymal hemorrhage (PH) (%) at day 1, the change on the NIHSS score from baseline to 1 day, the change on the NIHSS score from baseline to 7 day, mRS 0-1 (%) at 90 day, and mRS at 90 day.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with anterior circulation acute ischaemic stroke who are eligible for alteplase and mechanical thrombectomy commenced within 24 hours of stroke onset or awakening with stroke (if within 24 hours from the midpoint of sleep).
* Patient's age is 18-85 years.
* Arterial occlusion on CTA of the ICA, M1 or M2.
* Imaging inclusion criteria: infarct core volume ≤ 100 mL and penumbra ≥ 15 mL with at least 20% mismatch (as evaluated by CTP).
* Patient, family member or legally responsible person depending on local ethics requirements has given informed consent.

Exclusion Criteria:

* Pre-existing neurologic disability (a score greater than 2 on the mRS).
* Contraindication of fingolimod.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
independent recovery assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 (%) | at 90 day
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
salvaged ischemic tissue index (%) | from baseline to 7 day
  100*(baseline CTP ischemic lesion (mL) - 7 day DWI infarction lesion (mL))/ baseline CTP ischemic lesion (mL)
the growth in infarct volume (mL) | from 24 hour to 7 day
  24 hour DWI infarct volume (mL) - 7 day DWI infarct volume (mL)
the penumbral salvage volume (mL) | from baseline to 1 day
  (baseline CTP hypoperfusion volume (mL) - 24 hour DWI infarct volume (mL))
the frequency of parenchymal hemorrhage (PH) (%) | at day 1
  the presence of PH is defined according the standard from ECASS-2 study
the change on the National Institute of Health stroke scale (NIHSS) score from baseline to 1 day | from baseline to 1 day
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
the change on the National Institute of Health stroke scale (NIHSS) score from baseline to 7 day | from baseline to 7 day
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
excellent recovery assessed by the ratio of modefied Rankin Scale (mRS) score of 0-1 (%) | at day 90
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
general recovery assessed by the ratio of modefied Rankin Scale (mRS) score of 0-3 (%) | at day 90
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
recovery assessed by modefied Rankin Scale (mRS) score | at day 90
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, MD, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided